CLINICAL TRIAL: NCT00370825
Title: Combination Chemotherapy for the Treatment of Indian Visceral Leishmaniasis: Miltefosine Plus Liposomal Amphotericin B - Dose and Duration Ranging Study
Brief Title: Combination Chemotherapy for the Treatment of Indian Kala-Azar
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Banaras Hindu University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KAMRC0601
Record Dates: First submitted 2006-08-31; First posted 2006-09-01 (Estimated); Last update posted 2008-09-12 (Estimated); Status verified 2008-09

CONDITIONS: Visceral Leishmaniasis
Keywords: Visceral leishmaniasis; miltefosine; AmBisome; Combination
MeSH Terms: conditions — Leishmaniasis, Visceral | interventions — Combined Modality Therapy; liposomal amphotericin B; miltefosine

INTERVENTIONS:
Drug: Combination therapy with AmBisome and miltefosine

SUMMARY:
The investigators are using a sequential design to combine miltefosine and AmBisome in different doses.

DETAILED DESCRIPTION:
In this sequential design four arm study one arm is a reference arm but the three arms will consist an of initial dose of liposomal amphotericin B on first day followed by miltefosine. Both the drugs will be used in different doses. Reference arm will consist only a single dose of amBisome at 5 mg/kg. After the end of treatment, the post treatment assessment will be done on day 16 (initial cure) and six months (final cure). Safety parameters will be evaluated on day 0, 8 and 16. An arm with an efficacy of less than 75% will be closed. There will be periodical assessment of study results after completion of 5 patients in each arm.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of active VL with consistent signs and symptoms (e.g., fever, splenomegaly).
* Confirmed diagnosis by bone-marrow or splenic aspirate smear showing characteristic amastigotes.
* Male or female.
* Ages 12 to 65 years.
* Both newly diagnosed cases and patients who have received previous treatment (in the latter case a 2-week wash-out will be required before starting the study treatment).
* WBC > 1,000/mm3.
* Hemoglobin ≥ 4 g/dL

Exclusion Criteria:

* Pregnancy or breast-feeding.
* HIV positive serology.
* ASAT, ALAT, AP ≥ 3 times upper limit of normal range.
* Bilirubin ≥ 2 times upper limit of normal range.
* Prothrombin time ≥ 5 seconds above control.
* Serum creatinine or BUN ≥ 1.5 times upper limit of normal range.
* Any medical condition or situation that compromises compliance with study procedures.
* HIV

Ages: 12 Years to 65 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Enrollment: 200
Dates: Start 2006-09

PRIMARY OUTCOMES:
Absence of clinical kala-azar at six month follow up

CONTACTS AND LOCATIONS:
Overall Officials: Shyam Sundar, MD, Principal Investigator — Banaras Hindu University
Locations (1):
- Kala-azar Medical Research Center, Muzaffarpur, Bihar, India

REFERENCES:
- [Derived] Sundar S, Rai M, Chakravarty J, Agarwal D, Agrawal N, Vaillant M, Olliaro P, Murray HW. New treatment approach in Indian visceral leishmaniasis: single-dose liposomal amphotericin B followed by short-course oral miltefosine. Clin Infect Dis. 2008 Oct 15;47(8):1000-6. doi: 10.1086/591972. PMID 18781879